CLINICAL TRIAL: NCT00584883
Title: A Phase I Study of ABT 510 and Concurrent Temozolomide and Radiotherapy for Patients With Newly Diagnosed Glioblastoma Multiforme
Brief Title: A Phase I Study of ABT 510 for Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Louis Burt Nabors, MD, Professor, Neurology, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAB 0327; ABT510 (Other: Drug name from FDA)
Record Dates: First submitted 2007-12-26; First posted 2008-01-02 (Estimated); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Brain Tumor
Keywords: Patients who have newly diagnosed brain tumors
MeSH Terms: conditions — Brain Neoplasms | interventions — NAc-Sar-Gly-Val-(d-allo-Ile)-Thr-Nva-Ile-Arg-ProNEt

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ABT 510 (Experimental): The only arm will receive the ABT 510 following standard therapy with radiation and temozolomide chemotherapy concurrent.
  Interventions: Drug: ABT 510

INTERVENTIONS:
Drug: ABT 510 — ABT 510 (TSP-1 mimetic peptide) is a parenterally available nonapeptide analog of the heptapeptide and is a potent inhibitor of angiogenesis. ABT 510 competes with TSP-1 for binding to endothelial cells, but the exact mechanism of anti-angiogenesis is unknown. ABT 510 is administered by SQ injection. The starting dose of ABT 510 will be 20mg once daily (QD) SQ. Doses will be escalated by approximately 50% increments in consecutive cohorts of 3-6 patients until maximum tolerated dose is achieved.

SUMMARY:
To determine the maximum tolerated dose of ABT 510 when administered concurrent with radiation therapy for patients with newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
1. To describe the toxicity associated with this regimen in adult patients with newly diagnosed glioblastoma multiforme.
2. To determine the duration of disease free survival and overall survival associated with this therapy.
3. Evaluate thrombospondin 1 (TSP-1) and 2 (TSP-2) in tumor vs. corresponding normal tissue using quantitative real time Polymerase Chain Reaction (Q-RT-PCR).
4. Determine the effect of ABT 510 on tumor permeability and tumor blood volume as measured by non-invasive Magnetic Resonance Imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 19 years of age or older.
2. Patients must have histologically proven newly diagnosed glioblastoma multiforme.
3. Patients must have fully recovered from the immediate post-operative period and be maintained on a stable corticosteroid regimen for 5 days prior to entry.
4. Patients must have a Karnofsky performance status > 60% (i.e. the patient must be able to care for himself/herself with occasional help from others).
5. Patients must have adequate hematologic, renal and liver function (i.e. Absolute neutrophil count > 1500/mm3, Platelets > 100,000/mm3, creatinine 1.5 mg/dl .
6. Women of childbearing potential must have a negative pregnancy test.
7. Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. The effect of the investigational drugs on the developing human fetus is not known, but these drugs are likely to be harmful to the developing fetus or nursing infant. Women of child-bearing potential must agree to use adequate contraception (either surgical sterilization; approved hormonal contraceptives such as birth control pills Depo-Provera, or Lupron Depot; barrier methods such as condom or diaphragm along with spermicide; or an Intrauterine device (IUD)). Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician and study PI immediately.
8. The patient is able to self-administer or has a caregiver who can reliably administer subcutaneous injections.
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Pregnant or breast feeding.
2. Prior therapy for the brain tumor (except surgery)
3. Prior treatment with antineoplastic agents.
4. Exclude sexually active males and females unwilling to practice contraception during the study.
5. Serious concurrent infections.
6. Clinically significant cardiac disease not well controlled with medication (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias ) or myocardial infarction within the last 12 months.
7. Patients who have had prior cytotoxic chemotherapy prior to radiation therapy.
8. Patients with other serious uncontrolled co-morbid diseases that the investigator feels may comprise the study findings.
9. Patients must be able to learn to self -administer or have another person administer subcutaneous(SQ) injections.
10. Patients who have received any other investigational agents within the 28 days prior to Day 1 of the study.

    -

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
All patients enrolled in this study will be statistically characterized for baseline and disease characteristics using descriptive statistics for continuous measures. | up to 2 years
  The primary outcome for the study was safety and to define the MTD (max tolerated dose). Also, survival was to be measured but the study was not powered to statistically have significance for that measure.

CONTACTS AND LOCATIONS:
Overall Officials: Louis B Nabors, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States